CLINICAL TRIAL: NCT00913289
Title: Liver Regeneration Therapy Using Autologous Adipose Tissue Derived Stromal Cells
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Kanazawa University (Other)
Responsible Party: Principal Investigator, Shuichi Kaneko, Professor, Kanazawa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 675
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Liver Cirrhosis
Keywords: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

ARMS (1):
- adipose tissue derived stromal cells (Other)
  Interventions: Biological: adipose tissue derived stromal cells

INTERVENTIONS:
Biological: adipose tissue derived stromal cells — dosage

SUMMARY:
Mesenchymal stem cells have the capability to differentiate into hepatocytes and will be useful for liver regeneration. Adipose tissue is relatively enriched with mesenchymal stem cells compared to bone marrow tissue. In this trial, eligible liver cirrhosis patients will receive autologous adipose tissue derived stromal cells which include such mesenchymal stem cells.

DETAILED DESCRIPTION:
The population of the liver cirrhosis patients is enormous in Japan and the only radical treatment for them is liver transplantation. However, the number of giving donors is extremely limited. Mesenchymal stem cells have been capable to differentiate into mesodermal-lineage cells as well as endodermal-lineage cells such as hepatocytes. They reside in the mesenchymal tissues such as bone marrows as well as adipose tissues. The latter tissues are relatively enriched with mesenchymal stem cells compared to bone marrow cells. In this study, the cirrhotic patients will receive autologous adipose tissue derived stromal cells which contains substantial number of mesenchymal stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis patients
* Platelets count in peripheral blood: over 7.0x10^4/microliter
* Serum creatinine: less than 1.5 mg/dl
* Capable of understanding the features of this clinical trial

Exclusion Criteria:

* Associated with risky gastroesophageal varices for bleeding
* Severe portal hypertension
* Complicated with severe heart failure
* Renal disease
* Respiratory disease
* Hematological disease
* Coagulation disturbance and judged to be excluded by doctors
* Associated with malignancy
* Past history of the following:

  * malignancy
  * ischemic heart disease
  * cerebrovascular disease (cerebral infarction, cerebral hemorrhage)
  * decompensated status of liver cirrhosis
* Pregnant, or possibility of pregnancy
* Infected with HIV
* Under mediation with adrenal corticoid steroid, anti-histamine drug
* Anticipated with difficulty of follow-up observation
* Anticipated with inconsistency of following the protocol
* Addiction of alcohol drinking and unable to stop drinking
* Other candidates who are judged to be not applicable to this study by doctors

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
all cause harmful events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shuichi Kaneko, M.D., Study Chair — Kanazawa University
Locations (1):
- Kanazawa University Hospital, Kanazawa, Ishikawa-ken, Japan